CLINICAL TRIAL: NCT03792542
Title: Anlotinib Hydrochloride for Advanced Soft Tissue Sarcoma Patients Who do Not Receive Chemotherapy:a One-arm, Multi-center, Prospective Clinical Trial(ALTER-S003)
Brief Title: Anlotinib Hydrochloride For Advanced Soft Tissue Sarcoma Patients Who Do Not Receive Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Ningbo No.2 Hospital (Other); The Third People's Hospital of Hangzhou (Other); Jiangsu Provincial People's Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-S003
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib Hydrochloride ( 12mg, quaque die（QD）, PO, d1-14, 21 days per cycle), take once when limosis in the morning. If patients cannot suffer from adverse events(AEs), they can get declined dosage.
  Other Names: AL3818

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor. It can inhibit the angiogenesis related kinase, such as Vascular Endothelial Growth Factor Receptor (VEGFR), Fibroblast Growth Factor Receptor(FGFR), Platelet-Derived Growth Factor Receptor(PDGFR), and tumor cell proliferation related kinase c-Kit kinase. Anlotinib is an efficient second line therapeutic agent in treatment for metastatic soft tissue sarcoma which has been approved in clinical trials (ALTER-0203). There is a sort of patients who are not candidate for standard first line chemotherapy that is doxorubicin based. The patients either refused or too old and and debilitated to receive the cytotoxic chemotherapy.

DETAILED DESCRIPTION:
This study is planned to be carried out in Zhejiang and Jiangsu province regional multi-center. 44 cases are preliminarily expected to be included. The study started in January 2019 and ended in December 2019. It is expected that the trial will end in December 2020.

In the absence of such situations as withdrawal of informed consent, intolerance of drug toxicity and side effects, or inappropriateness for further trials, each participant's expected time for research and treatment will continue until radiographically confirmed tumor progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to patient entry;
* ≥ 18 and ≤ 70 years of age , regardless of gender；ECOG :0-2;Expected Survival Time: Over 3 months;
* Histologically confirmed diagnosis of un-resectable or recurrent metastatic soft tissue sarcoma, such as: leiomyosarcoma, synovial sarcoma, undifferentiated pleomorphic sarcoma, liposarcoma and other sarcomas. The following histologies are excluded: alveolar Soft tissue sarcoma, rhabdomyosarcoma, chondrosarcoma, osteosarcoma, gastrointestinal stromal tumor, humeral cutaneous fibrosarcoma, Ewing sarcoma/primary neuroectodermal tumor, inflammatory myofibroblastic sarcoma and malignant mesothelioma.
* Patients who have not treated with anti-tumor drugs, or it has been more than 6 months after the end of adjuvant and neoadjuvant chemotherapy.
* Refuse the firs-line chemotherapy or could not tolerate chemotherapy as determined by treatment physician
* Evaluable disease by imaging or physical exam or measurable disease defined as at least one lesion that can be accurately measured according to RECIST version 1.1.
* normal main organs function as defined below: Hemoglobin (Hb) ≥ 80g / L, Neutrophils (ANC) ≥ 1.5 × 109 / L, Platelet count (PLT) ≥ 80 × 109 / L, Serum creatinine (Cr) ≤ 1.5 × normal upper limit (ULN) or creatinine clearance (CCr) ≥ 60ml / min, Blood urea nitrogen (BUN) ≤ 2.5 × normal upper limit (ULN); Total bilirubin (TB) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; If accompanied by liver metastases, ALT and AST ≤ 5 × ULN Albumin (ALB) ≥ 25 g/L. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%)
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped.

Exclusion Criteria:

* Appropriate and willing for cytotoxic chemotherapy.
* Prior systemic therapy for this type of sarcoma. Neoadjuvant or adjuvant therapy more than 6 months prior would not apply.
* Prior treatment with any VEGFR tyrosine kinase inhibitor(such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib, apatinib, regorafenib and other drugs).
* Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy, is planned for the first 4 weeks prior to enrollment or during the study. Radiation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
* A history of other malignancy ≤ 5 years previous with the exception of cured cervical carcinoma in situ, cutaneous basal cell carcinoma or squamous cell carcinoma of the skin.
* Known brain metastases.
* The investigator judged that during the follow-up study, the tumor is very likely to invade the important blood vessels and cause fatal hemorrhage, or the formation of tumor thrombosis with large veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava);
* unable to swallow and retain oral capsules.
* with any severe and/or uncontrolled disease, including:1)Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment).2)Arrhythmias with grade II and above myocardial ischemia or myocardial infarction, poor control (including corrected QT interval(QTc) men ≥ 450 ms, women ≥ 470 ms) and ≥ 2 congestive heart failure (New York Heart Association ( NYHA) rating).3)Poor control of diabetes (fasting blood glucose > 10mmol / L).4)Active or uncontrolled serious infection (≥ Common Terminology Criteria for Adverse Event(CTC AE) grade 2 infection);5)Patients with active hepatitis B or hepatitis C (hepatitis B: HBsAg-positive and hepatitis B virus(HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus(HCV) RNA-positive and abnormal liver function), or active infection requiring antimicrobial treatment (eg Treated with antibacterial drugs, antiviral drugs, antifungal drugs);6)renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;7)Patients with seizures and need treatment
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time(APTT) > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy.
* Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin.
* significant coughing blood in the 2 months before enrollment, or daily hemoptysis of 2.5ml or more.
* history of psychotropic substance abuse who are unable to quit or have a mental disorder.
* Tendencies of hereditary or acquired hemorrhagic and thrombotic (such as hemophilia patients, coagulopathy, thrombocytopenia, hypersplenism, etc.)
* Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks and/or had any bleeding or bleeding episodes which the degree is bigger than CTCAE 3 grade within 4 weeks prior to enrollment.
* Active period digestive ulcers.
* Cavity sinus or perforation occurred within 6 months.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Received a potent CYP3A4 inhibitor (such as ketoconazole, itraconazole, erythromycin, and clarithromycin) within 7 days, or received a potent CYP3A4 inducer within 12 days prior to the study (eg. catarrh Treatment with imipramine, rifampicin and phenobarbital).
* Allergic reactions, hypersensitivity reactions or intolerance to anlotinib hydrochloride or its excipients.
* Pregnancy or lactation.
* The investigator believes that there are any conditions that may damage the subject or result in the subject not being able to meet or perform the research request.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | until Progressive Disease(PD) or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Quality of Life score (QoL) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoming Ye, professor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China